CLINICAL TRIAL: NCT05106296
Title: Repurposing Ibrutinib for Chemo-Immunotherapy in a Phase 1b Study of Ibrutinib With Indoximod Plus Metronomic Cyclophosphamide and Etoposide for Pediatric Patients With Brain Cancer
Brief Title: Chemo-immunotherapy Using Ibrutinib Plus Indoximod for Patients With Pediatric Brain Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Theodore S. Johnson (Other)
Collaborators: Augusta University (Other); CureSearch for Children's Cancer (Unknown); Rally Foundation for Childhood Cancer Research (Other)
Responsible Party: Sponsor-Investigator, Theodore S. Johnson, Professor of Pediatrics and Co-Director of the Pediatric Immunotherapy Program, Augusta University
Organization: Augusta University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCC2020
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Ependymoma; Medulloblastoma; Glioblastoma; Primary Brain Tumor
Keywords: IDO; indoleamine 2,3-dioxygenase; indoximod; BTK; Bruton's Tyrosine Kinase; ibrutinib; immunotherapy; pediatric; childhood; brain tumor; brain cancer; glioblastoma; medulloblastoma; ependymoma; PNET; cyclophosphamide; etoposide; immune; central nervous system; CNS; temozolomide
MeSH Terms: conditions — Ependymoma; Medulloblastoma; Glioblastoma; Brain Neoplasms; Neuroectodermal Tumors, Primitive | interventions — 1-methyltryptophan; ibrutinib; Cyclophosphamide; Etoposide; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Regimen A (Experimental): Patients will be treated with ibrutinib plus indoximod, cyclophosphamide, and etoposide. Cycles are a minimum of 28 days.
  Interventions: Drug: Indoximod; Drug: Ibrutinib; Drug: Cyclophosphamide; Drug: Etoposide
- Regimen B (Experimental): Patients will be treated with ibrutinib plus indoximod and temozolomide. Cycles are a minimum of 28 days.
  Interventions: Drug: Indoximod; Drug: Ibrutinib; Drug: Temozolomide

INTERVENTIONS:
Drug: Indoximod — Indoximod will be taken by mouth twice daily, throughout each treatment cycle.
Drug: Ibrutinib — For Regimen A, Ibrutinib will be taken by mouth once daily, on days 1-21 of each treatment cycle.
  Arms: Regimen A
Drug: Cyclophosphamide — Cyclophosphamide will be taken by mouth once daily, on days 1-21 of each treatment cycle.
  Arms: Regimen A
Drug: Etoposide — Etoposide will be taken by mouth once daily, on days 1-21 of each treatment cycle.
  Arms: Regimen A
Drug: Ibrutinib — For Regimen B, Ibrutinib will be taken by mouth once daily, on days 1-14 of each treatment cycle.
  Arms: Regimen B
Drug: Temozolomide — Temozolomide will be taken by mouth once daily, on days 1-5 of each treatment cycle.
  Arms: Regimen B

SUMMARY:
Recent lab-based discoveries suggest that IDO (indoleamine 2,3-dioxygenase) and BTK (Bruton's tyrosine Kinase) form a closely linked metabolic checkpoint in tumor-associated antigen-presenting cells. The central clinical hypothesis for the GCC2020 study is that combining ibrutinib (BTK-inhibitor) with indoximod (IDO-inhibitor) during chemotherapy will synergistically enhance anti-tumor immune responses, leading to improvement in clinical response with manageable overlapping toxicity.

The GCC2020 trial is a prospective open-label phase 1 trial to determine the best safe dose of the BTK-inhibitor ibrutinib to use in combination with previously studied chemo-immunotherapy regimens comprised of the investigational IDO-inhibitor indoximod plus oral palliative chemotherapy for participants, age 6 to 25 years, with relapsed or refractory primary brain cancer. Those previously treated with indoximod-based therapy may be eligible, including prior treatment via the phase 2 indoximod study (GCC1949, NCT04049669), the now closed phase 1 study (NLG2105, NCT02502708), or any expanded access (compassionate use) protocols. Ibrutinib will be combined with either indoximod plus oral cyclophosphamide and etoposide (Regimen A) or indoximod plus oral temozolomide (Regimen B). No cross-over between these two regimens will be allowed. Dose-escalation cohorts will determine the best safe dose of ibrutinib for each of these regimens. This will be followed by expansion cohorts, using ibrutinib at the best safe dose for each regimen, to allow assessment of preliminary evidence of efficacy.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis:

* Patients must have prior documented progressive or refractory disease with histologically proven initial diagnosis of ependymoma, medulloblastoma, glioblastoma, or another type of primary cancer of the central nervous system with no curative conventional therapy options available.
* Metastatic disease is acceptable.
* Patients must have MRI confirmation (with and without gadolinium contrast) of current active disease.

Patients must be able to swallow pills.

Lansky or Karnofsky performance status score must be ≥ 50%.

Adequate renal function:

* Creatinine clearance (CLcr) > 25 mL/min (by calculated methods) AND Creatinine ≤ 1.5-times upper limit of age-adjusted normal for age of patient.

Adequate liver function:

* Alanine aminotransferase (ALT) ≤ 3-times upper limit of normal.
* Aspartate aminotransferase (AST) ≤ 3-times upper limit of normal.
* Total bilirubin ≤ 1.5-times upper limit of normal unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin.

Adequate bone marrow function:

* Absolute neutrophil count (ANC) ≥ 1000/mm3 (independent of growth factor support).
* Platelets ≥ 100,000/mm3 (independent of transfusion support).
* Hemoglobin ≥ 8 g/dL (independent of transfusion support).

Seizure disorders must be well controlled on antiepileptic medication.

Prior therapy:

* Patients previously treated with chemotherapy drugs included in this protocol are eligible for enrollment.
* At the time of Screening, patients must be at least 21 days from the administration of any investigational agent (other than indoximod) or prior cytotoxic therapy (including chemotherapy).
* At the time of Screening, patients must be at least 28 days from administration of antibody-based therapies (e.g., bevacizumab), tumor-directed vaccines, or cellular immune therapies (e.g., T cells, NK cells, etc.).
* At the time of Screening, patients must be at least 56 days from administration of tumor-directed therapies using infectious agents (e.g., viruses, bacteria, etc.).
* At the time of Screening, patients must be at least 90 days from any radiation or proton therapy (all modalities, including radiosurgery) that targeted all sites of known disease.
* There is no lock-out window for patients who were treated with focal radiation or focal proton therapy (all modalities, including radiosurgery) that did not target all disease sites, if at least one site of active tumor is expected to persist and/or grow.

Concurrent anti-neoplastic therapy:

* No investigational or commercial agents, including intrathecal drugs, other than that described by this clinical study protocol (GCC2020) may be administered with the intent to treat the patient's malignancy while they remain enrolled on this study.

Contraception, pregnancy, and breastfeeding:

* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study. Men must agree to not donate sperm during and for 3 months after the study.
* Women who are pregnant or breastfeeding are ineligible for this study.
* Patients who become pregnant while participating in this study will have to stop Study Therapy.

Patients, or their parent for patients less than 18 years of age, must sign an Informed Consent Document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study.

.

Exclusion Criteria:

Patients who are unable to swallow pills.

Patients with known hypersensitivity to any drugs in the treatment plan.

Patients with active autoimmune disease that requires systemic therapy.

* Allergies, allergic conditions, and reactive inflammatory conditions that are not autoimmune in nature would not exclude patients (e.g., eczema, asthma, etc.).

Pregnant or breastfeeding women.

Major surgery or a wound that has not fully healed within 4 weeks of Screening.

Known central nervous system lymphoma.

Patients with active bleeding or history of thrombotic or hemorrhagic stroke, or intracranial hemorrhage, within 6 months prior to Screening; with the exception of retained blood products from recent prior uncomplicated surgery (e.g., tumor biopsy, debulking, or resection; VP shunt placement, etc.).

Requires anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon).

Requires chronic treatment with strong CYP3A inhibitor drugs.

Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.

Patients with baseline QTc interval of more than 470 msec at the time of Screening, and patients with congenital long QT syndrome.

Vaccinated with live, attenuated vaccines within 4 weeks of Screening.

Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection.

Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of ibrutinib, indoximod, or chemotherapy, or put the study outcomes at undue risk.

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-02-08 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of regimen-limiting toxicity (RLT) for Regimen A | First 90 days of treatment
  To determine the pediatric recommended phase 2 dose (RP2D) of ibrutinib, when combined with indoximod-based chemo-immunotherapy (Regimen A)
Objective Response Rate (ORR) for Regimen A | Up to 5 years
  Defined as the proportion of patients with a best objective response of either complete response (CR) or partial response (PR), using "immunotherapy Response Assessment for Neuro-Oncology" (iRANO) criteria
Incidence of regimen-limiting toxicity (RLT) for Regimen B | First 90 days of treatment
  To determine the pediatric recommended phase 2 dose (RP2D) of ibrutinib, when combined with indoximod-based chemo-immunotherapy (Regimen B)
Objective Response Rate (ORR) for Regimen B | Up to 5 years
  Defined as the proportion of patients with a best objective response of either complete response (CR) or partial response (PR), using "immunotherapy Response Assessment for Neuro-Oncology" (iRANO) criteria

SECONDARY OUTCOMES:
Adverse events (AEs) | Up to 19 months
  To assess frequency, severity, and recoverability of AEs for the treatment regimen
Frequency of cycle delays for toxicity | Up to 18 months
  To assess whether the immunotherapy contributes to delays in starting subsequent cycles of the chemotherapy drugs
Frequency of dose-reductions of the chemotherapy regimen | Up to 18 months
  To assess whether the immunotherapy contributes to reductions in the doses of the chemotherapy drugs
Complete Response Rate (CRR) | Up to 5 years
  Defined as the proportion of patients with a best objective response of CR using iRANO criteria
Partial Response Rate (PRR) | Up to 5 years
  Defined as the proportion of patients with a best objective response of PR using iRANO criteria
Modified Objective Response Rate (mORR) | Up to 5 years
  Defined as the proportion of patients with best objective response of complete response (CR), partial response (PR), or stable disease (SD, on at least 2 sequential study-timed MRIs) using iRANO criteria
iRANO-PFS | Up to 5 years
  Time of Progression-Free Survival (PFS), defined as time from study entry to progression using iRANO criteria
Overall Survival (OS) | Up to 5 years
  Time from study entry to death

CONTACTS AND LOCATIONS:
Overall Officials: Theodore S. Johnson, MD, PhD, Principal Investigator — Augusta University
Locations (1):
- Augusta University, Georgia Cancer Center, Augusta, Georgia, United States

REFERENCES:
- [Background] Johnson TS, MacDonald TJ, Pacholczyk R, Aguilera D, Al-Basheer A, Bajaj M, Bandopadhayay P, Berrong Z, Bouffet E, Castellino RC, Dorris K, Eaton BR, Esiashvili N, Fangusaro JR, Foreman N, Fridlyand D, Giller C, Heger IM, Huang C, Kadom N, Kennedy EP, Manoharan N, Martin W, McDonough C, Parker RS, Ramaswamy V, Ring E, Rojiani A, Sadek RF, Satpathy S, Schniederjan M, Smith A, Smith C, Thomas BE, Vaizer R, Yeo KK, Bhasin MK, Munn DH. Indoximod-based chemo-immunotherapy for pediatric brain tumors: A first-in-children phase I trial. Neuro Oncol. 2024 Feb 2;26(2):348-361. doi: 10.1093/neuonc/noad174. PMID 37715730
- [Background] Sharma MD, Pacholczyk R, Shi H, Berrong ZJ, Zakharia Y, Greco A, Chang CS, Eathiraj S, Kennedy E, Cash T, Bollag RJ, Kolhe R, Sadek R, McGaha TL, Rodriguez P, Mandula J, Blazar BR, Johnson TS, Munn DH. Inhibition of the BTK-IDO-mTOR axis promotes differentiation of monocyte-lineage dendritic cells and enhances anti-tumor T cell immunity. Immunity. 2021 Oct 12;54(10):2354-2371.e8. doi: 10.1016/j.immuni.2021.09.005. Epub 2021 Oct 5. PMID 34614413